CLINICAL TRIAL: NCT01246089
Title: Ranibizumabe Intravitreal Injection for Myopic Choroidal Neovascularization
Brief Title: Ranibizumab for Myopic Neovascularization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, MD, Instituto de Olhos de Goiania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JN-09-2010-AR
Record Dates: First submitted 2010-11-20; First posted 2010-11-23 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Myopic Choroidal Neovascularization
Keywords: Ranibizumab; Myopia; Complications; Neovascularization; OCT
MeSH Terms: conditions — Myopia; Neovascularization, Pathologic | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranabizumab (Experimental): Myopic eyes with retinal neovascularization
  Interventions: Drug: ranibizumab injection

INTERVENTIONS:
Drug: ranibizumab injection — Ranibizumab intravitreal injection of 0,5 mg ( 0.05mL)

SUMMARY:
The purpose of this study is to evaluate the clinical results of anti-VEGF intra-vitreal injections (IVT) in CNV secondary to pathologic myopia (PM-CNV).

DETAILED DESCRIPTION:
Twenty consecutive patients (30 eyes) with subfoveal PM-CNV, 9 of whom had been unsuccessfully treated with Visudyne PDT, were treated with IVT of 0.5mg ranibizumab. ETDRS best corrected visual acuity, macular thickness on OCT scans, and angiographic features were recorded and evaluated. The aspect of OCT scans passing across the PM-CNV was also analyzed. IVTs were repeated only in case of persistent angiographic leakage and if OCT scans showed retinal thickening or edema and serous retinal detachment. The follow-up period was at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Myopic and CNVM

Exclusion Criteria:

* Patients with poor compliance

  * Patients with uncontrolled diabetes and hypertension or any other medical condition that increase the risk of complications like recent history of Stroke or myocardial infraction (< one year). (Physician clearance was obtained for all patients).
  * Age related macular degeneration with Juxtafoveal and Subfoveal CNVM: Recurrent CNVM following PDT and TTT with IVTA. Patient who could not afford PDT, Macugen or Lucentis which is FDA approved.
  * Patients who had undergone major surgery 28 days before, were excluded from the study and it was also suspended prior to elective surgery.
  * Refractory macular oedema due to vein occlusion, Pseudophakia, Clinically significant macular oedema (CSME) etc. that affects vision and does not respond adequately to usual treatment methods.
  * Proliferative diabetic retinopathy, non-resolving vitreous haemorrhage with PDR.
  * Idiopathic CNVM, Inflammatory CNVM and other conditions associated with CNVM.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil